CLINICAL TRIAL: NCT02185781
Title: Phase I Protocol of Adoptive Immunotherapy With Enriched and Expanded Autologous Natural Killer (NK) Cells for Patients With Ph+ Acute Lymphoblastic Leukemia (ALL) in Complete Hematologic Remission (CHR) But With Persistent/Recurrent Minimal Residual Disease (MRD) ≥60 Years or Not Eligible for Other Post-CHR Treatment Modalities
Brief Title: Phase I Study of Adoptive Immunotherapy With Enriched and Expanded Autologous Natural Killer (NK) Cells for Patients With Ph+ Acute Lymphoblastic Leukemia (ALL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL 2013
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Acute Lymphoblastic Leukemia; Complete Hematologic Remission (CHR); Persistent/Recurrent Minimal Residual Disease (MRD)
Keywords: Phase I; Adoptive immunotherapy; Enriched and expanded autologous natural killer (NK) cells; Ph+ acute lymphoblastic leukemia; ≥60 years; Not eligible for other post-CHR treatment modalities
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous NK Cells infusions (Experimental)
  Interventions: Other: Autologous NK cells infusions

INTERVENTIONS:
Other: Autologous NK cells infusions — Each patient will receive repeated intravenous (IV) infusions of escalating doses of expanded autologous NK cells.
  The initial dose will be 1 x 106/kg of recipient body weight (BW), followed by half log increments of the dose level for each infusion, to a maximum of 1 x 108/kg of recipient BW or until they experience any toxicity, for a maximum of 5 infusions. The minimum interval between each infusion will be 28 days. No conditioning therapies will be administered before the infusion of the expanded NK cells. Patients may receive TKI maintenance.

SUMMARY:
The present study aims at studying how safe and tolerable a new therapy for patients with Acute Lymphoblastic Leukemia (ALL) is.

This new therapy consists of an immunotherapy, that is an approach focusing on the immune system, and it targets ALL patients in complete remission but who may still have the disease at a cellular level (this is called 'minimal residual disease').

For any further information, please, discuss with your treating physician.

DETAILED DESCRIPTION:
This is an open label, multicenter, phase I study of adoptive immunotherapy with enriched and expanded autologous natural killer (NK) cells for patients with Ph+ acute lymphoblastic leukemia (ALL) in complete hematologic remission (CHR) but with persistent/recurrent minimal residual disease (MRD) ≥60 years or not eligible for other post-CHR treatment modalities.

The study will investigate the safety and tolerability of a new type of NK-based immunotherapy based on the infusion of escalating doses of ex-vivo expanded autologous NK cells in Ph+ ALL patients. A maximum of 6 patients will be enrolled in two different steps. No conditioning therapies will be administered before the infusion of the expanded NK cells. Patients may receive tyrosine kinase inhibitor (TKI) maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with Ph+ ALL in CHR (1st or 2nd) with MRD positivity confirmed at baseline, older or equal to 60 years or not eligible for other post-CHR treatment modalities.
* WHO score 0-1.
* Hematopoietic, liver and renal normal functions defined as follows:

WBC bigger or equal to 2.000/mm3 lymphocytes bigger or equal to 500/mm3 neutrophils bigger or equal to 1.000/mm3 platelets bigger or equal to 50.000/mm3 Hb bigger or equal to 9 g/dl creatinine fewer or equal to 1.5 x ULN bilirubin fewer or equal to 1.5 x ULN AST and ALT less than 3 times the upper limit of normal. LDH less than 2 times the upper limit of normal.

* For male and female subjects of childbearing potential, agreement to use effective contraception.
* Authorization by Istituto Superiore di Sanità (ISS) according to DM 2 March 2004.
* Signed written informed consent according to ICH/EU/GCP and national local regulations.

Exclusion Criteria:

* Concurrent chemotherapy or immunotherapy (TKI maintenance is permitted).
* Any contraindications to perform a leukapheretic procedure for mononuclear cell collection.
* Active or chronic infection, including Treponema, HIV, HBV and/or HCV unless antigen/PCR negative.
* Presence of autoimmune symptoms.
* Pregnant or lactating females.
* Simultaneous participation in another clinical trial.
* Any physical or psychological impediment in a patient that could lead the investigator to suspect his/her poor compliance to the protocol.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-01-28 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
To determine the MTD and the recommended final dose (RD) to be used for further investigations. | One year from start of treatment.

SECONDARY OUTCOMES:
Number of adverse events. | Two years from start of treatment.
  To assess the safety and tolerabilty of the treatment by evaluating frequency, type and intensity of adverse events (AEs) according to the CTC classification, as well as the patients' compliance and clinically relevant changes in the laboratory parameters.
Number of patients able to complete the study. | One year from start of treatment.
  To evaluate the feasibility of the procedure in terms of number of patients able to complete the study and time to complete enrolment.
Time to complete enrolment. | Three years from first patient enrollment.
  Protocol feasibility.
Number and characteristics of immunologic modifications. | One year from start of treatment.
  To assess the immunologic modifications induced by the procedure; in particular, to verify the functional and cytotoxic activity against tumor cell lines and primary fresh allogeneic and autologous blasts cryopreserved at diagnosis, and to monitor the frequency, phenotype and activation status of the infused NK cell populations by flow cytometry analyses, Chromium release cytotoxic assays and intracellular cytokine production.
Number of patients who respond to treatment. | One year from treatment start.
  To evaluate the clinical response to the treatment in terms of control of MRD with quantitative (Q)- RT-PCR.
Number of patients alive after treatment conclusion. | Two years from treatment start.
  To evaluate OS in terms of number of patients alive.
Number of patients alive without progression. | One year from treatment start.
  To evaluate the TTP in terms of number of patients alive without progression.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Foà, Study Chair — Policlinico Umberto I di Roma; Giovanni Torelli, Study Director — Policlinico Umberto I di Roma
Locations (6):
- Italy (6):
  - ISS/AIFA, Roma
  - Ospedale S. Eugenio, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - Università degli Studi - Policlinico di Tor Vergata, Roma
  - Università Degli Studi Di Roma "Sapienza" - Dipartimento Di Medicina Traslazionale E Di Precisione - U.O.C. Ematologia, Roma